CLINICAL TRIAL: NCT02988544
Title: Artificial Shrinkage of Fresh Blastocyst: Impact on Success Rates in Assisted Reproductive Technology
Brief Title: Artificial Shrinkage of Fresh Blastocysts
Acronym: BlastoCollapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RECHMPL16_0267
Record Dates: First submitted 2016-12-02; First posted 2016-12-09 (Estimated); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Infertility Assisted Reproductive Technology
Keywords: Single blastocyst embryo transfer; Artificial Shrinkage; Clinical pregnancy rate; Cell free

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artificial shrinkage (AS) group (Experimental): The Artificial shrinkage group where blastocoelic cavity is artificially reduced by a laser pulse prior to transfer
  Interventions: Procedure: Artificial shrinkage
- Control group (No Intervention): No intervention on blastocoelic

INTERVENTIONS:
Procedure: Artificial shrinkage — Artificial shrinkage of blastocyst
  Arms: Artificial shrinkage (AS) group

SUMMARY:
The aim of the study is to determine if collapsing an embryo (or making it fold compactly by taking away its fluid) before the transfer in the uterine cavity improves pregnancy rates in assisted reproductive technology (ART).

Women coming to our ART center will be randomized in two groups : the collapsing group and a control group.

Pregnancy rates will be compared in the two groups. A biomarker (cell free DNA) will also be determined in each group and correlated to pregnancy occurrence.

DETAILED DESCRIPTION:
This is a prospective randomized study designed to determine if artificial shrinkage (AS) before transfer of embryos impact clinical pregnancy rate in single blastocyst embryo transfer (SBET) cycle. Women elected for SBET will be randomized on transfer day in two arms:the AS group where blastocoelic cavity is artificially reduced by a laser pulse prior to transfer and a control group.

Clinical pregnancy rates will be compared. Secondarily, rate of monozygotic twin pregnancy and cell free DNA concentration in culture medium will be evaluated in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Couple eligible for a transfer of a single embryo at the blastocyst stage
* Available couple for a follow up of 12 months

Exclusion Criteria:

* Attempt with frozen embryo or frozen oocyte
* Attempt with a pre-implantation diagnosis
* Patient has not signed informed consent
* Couple in a period of exclusion determined by a previous study
* Couple under legal protection, guardianship or guardianship

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2018-05-20 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate embryo transfer | 5 weeks
  Clinical pregnancy rate by transfer evaluate by the visualization of at least one gestational sac with fetal heart activity during pelvic ultrasound confirmed by a positive result of the quantitative βHCG blood test.

SECONDARY OUTCOMES:
Twin pregnancy rate by transfer | 5 weeks
  Twin pregnancy rate by transfer evaluate the presence of 2 cardiac activities on ultrasound.
Free DNA level | Baseline
  Free DNA content contained in the drop of culture medium collected after transfer.

CONTACTS AND LOCATIONS:
Overall Officials: Anna AG GALA, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Montpellier University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Czamanski-Cohen J, Sarid O, Cwikel J, Lunenfeld E, Douvdevani A, Levitas E, Har-Vardi I. Increased plasma cell-free DNA is associated with low pregnancy rates among women undergoing IVF-embryo transfer. Reprod Biomed Online. 2013 Jan;26(1):36-41. doi: 10.1016/j.rbmo.2012.09.018. Epub 2012 Oct 4. PMID 23182744
- [Background] D'Alessandro A, Federica G, Palini S, Bulletti C, Zolla L. A mass spectrometry-based targeted metabolomics strategy of human blastocoele fluid: a promising tool in fertility research. Mol Biosyst. 2012 Apr;8(4):953-8. doi: 10.1039/c1mb05358b. Epub 2011 Oct 21. PMID 22020776
- [Background] Fanchin R, Ayoubi JM. Uterine dynamics: impact on the human reproduction process. Reprod Biomed Online. 2009;18 Suppl 2:57-62. doi: 10.1016/s1472-6483(10)60450-6. PMID 19406033
- [Background] Gala A, Ferrieres A, Assou S, Monforte M, Bringer-Deutsch S, Vintejoux E, Vincens C, Brunet C, Hamamah S. [Effects of artificial shrinkage prior to vitrification in a closed system: a randomized controlled trial]. Gynecol Obstet Fertil. 2014 Nov;42(11):772-8. doi: 10.1016/j.gyobfe.2014.09.006. Epub 2014 Oct 16. French. PMID 25442824
- [Background] Gianaroli L, Magli MC, Pomante A, Crivello AM, Cafueri G, Valerio M, Ferraretti AP. Blastocentesis: a source of DNA for preimplantation genetic testing. Results from a pilot study. Fertil Steril. 2014 Dec;102(6):1692-9.e6. doi: 10.1016/j.fertnstert.2014.08.021. Epub 2014 Sep 23. PMID 25256935
- [Background] Hammadeh ME, Fischer-Hammadeh C, Ali KR. Assisted hatching in assisted reproduction: a state of the art. J Assist Reprod Genet. 2011 Feb;28(2):119-28. doi: 10.1007/s10815-010-9495-3. Epub 2010 Nov 2. PMID 21042844
- [Background] Hur YS, Park JH, Ryu EK, Yoon HJ, Yoon SH, Hur CY, Lee WD, Lim JH. Effect of artificial shrinkage on clinical outcome in fresh blastocyst transfer cycles. Clin Exp Reprod Med. 2011 Jun;38(2):87-92. doi: 10.5653/cerm.2011.38.2.87. Epub 2011 Jun 30. PMID 22384424
- [Background] Iwayama H, Hochi S, Yamashita M. In vitro and in vivo viability of human blastocysts collapsed by laser pulse or osmotic shock prior to vitrification. J Assist Reprod Genet. 2011 Apr;28(4):355-61. doi: 10.1007/s10815-010-9522-4. Epub 2010 Dec 9. PMID 21152966
- [Background] Kato S, Janku F. Cell-free DNA as a novel marker in cancer therapy. Biomark Med. 2015;9(7):703-12. doi: 10.2217/bmm.15.38. PMID 26174844
- [Background] Kawachiya S, Bodri D, Shimada N, Kato K, Takehara Y, Kato O. Blastocyst culture is associated with an elevated incidence of monozygotic twinning after single embryo transfer. Fertil Steril. 2011 May;95(6):2140-2. doi: 10.1016/j.fertnstert.2010.12.018. Epub 2011 Jan 7. PMID 21215395
- [Background] Khalaf Y, El-Toukhy T, Coomarasamy A, Kamal A, Bolton V, Braude P. Selective single blastocyst transfer reduces the multiple pregnancy rate and increases pregnancy rates: a pre- and postintervention study. BJOG. 2008 Feb;115(3):385-90. doi: 10.1111/j.1471-0528.2007.01584.x. PMID 18190376
- [Background] Magli MC, Gianaroli L, Ferraretti AP. Chromosomal abnormalities in embryos. Mol Cell Endocrinol. 2001 Oct 22;183 Suppl 1:S29-34. doi: 10.1016/s0303-7207(01)00574-3. PMID 11576729
- [Background] MANDEL P, METAIS P. [Nuclear Acids In Human Blood Plasma]. C R Seances Soc Biol Fil. 1948 Feb;142(3-4):241-3. No abstract available. French. PMID 18875018
- [Background] Palini S, Galluzzi L, De Stefani S, Bianchi M, Wells D, Magnani M, Bulletti C. Genomic DNA in human blastocoele fluid. Reprod Biomed Online. 2013 Jun;26(6):603-10. doi: 10.1016/j.rbmo.2013.02.012. Epub 2013 Mar 13. PMID 23557766
- [Background] Scalici E, Traver S, Molinari N, Mullet T, Monforte M, Vintejoux E, Hamamah S. Cell-free DNA in human follicular fluid as a biomarker of embryo quality. Hum Reprod. 2014 Dec;29(12):2661-9. doi: 10.1093/humrep/deu238. Epub 2014 Sep 29. PMID 25267787
- [Background] Schieve LA, Meikle SF, Peterson HB, Jeng G, Burnett NM, Wilcox LS. Does assisted hatching pose a risk for monozygotic twinning in pregnancies conceived through in vitro fertilization? Fertil Steril. 2000 Aug;74(2):288-94. doi: 10.1016/s0015-0282(00)00602-6. PMID 10927046
- [Background] Schwarzenbach H, Hoon DS, Pantel K. Cell-free nucleic acids as biomarkers in cancer patients. Nat Rev Cancer. 2011 Jun;11(6):426-37. doi: 10.1038/nrc3066. Epub 2011 May 12. PMID 21562580
- [Background] Sharma VK, Vouros P, Glick J. Mass spectrometric based analysis, characterization and applications of circulating cell free DNA isolated from human body fluids. Int J Mass Spectrom. 2011 Jul;304(2-3):172-183. doi: 10.1016/j.ijms.2010.10.003. PMID 21765648
- [Background] Son WY, Yoon SH, Yoon HJ, Lee SM, Lim JH. Pregnancy outcome following transfer of human blastocysts vitrified on electron microscopy grids after induced collapse of the blastocoele. Hum Reprod. 2003 Jan;18(1):137-9. doi: 10.1093/humrep/deg029. PMID 12525454
- [Background] Stigliani S, Anserini P, Venturini PL, Scaruffi P. Mitochondrial DNA content in embryo culture medium is significantly associated with human embryo fragmentation. Hum Reprod. 2013 Oct;28(10):2652-60. doi: 10.1093/humrep/det314. Epub 2013 Jul 25. PMID 23887072
- [Background] Stigliani S, Persico L, Lagazio C, Anserini P, Venturini PL, Scaruffi P. Mitochondrial DNA in Day 3 embryo culture medium is a novel, non-invasive biomarker of blastocyst potential and implantation outcome. Mol Hum Reprod. 2014 Dec;20(12):1238-46. doi: 10.1093/molehr/gau086. Epub 2014 Sep 17. PMID 25232043
- [Background] Traver S, Scalici E, Mullet T, Molinari N, Vincens C, Anahory T, Hamamah S. Cell-free DNA in Human Follicular Microenvironment: New Prognostic Biomarker to Predict in vitro Fertilization Outcomes. PLoS One. 2015 Aug 19;10(8):e0136172. doi: 10.1371/journal.pone.0136172. eCollection 2015. PMID 26288130
- [Background] Van Landuyt L, Polyzos NP, De Munck N, Blockeel C, Van de Velde H, Verheyen G. A prospective randomized controlled trial investigating the effect of artificial shrinkage (collapse) on the implantation potential of vitrified blastocysts. Hum Reprod. 2015 Nov;30(11):2509-18. doi: 10.1093/humrep/dev218. Epub 2015 Sep 12. PMID 26364080
- [Background] Vanderzwalmen P, Bertin G, Debauche Ch, Standaert V, van Roosendaal E, Vandervorst M, Bollen N, Zech H, Mukaida T, Takahashi K, Schoysman R. Births after vitrification at morula and blastocyst stages: effect of artificial reduction of the blastocoelic cavity before vitrification. Hum Reprod. 2002 Mar;17(3):744-51. doi: 10.1093/humrep/17.3.744. PMID 11870130
- [Background] Warton K, Samimi G. Methylation of cell-free circulating DNA in the diagnosis of cancer. Front Mol Biosci. 2015 Apr 22;2:13. doi: 10.3389/fmolb.2015.00013. eCollection 2015. PMID 25988180
- [Background] Wu CL, Li HG, Zhu CH. [Advances in the studies of cell-free seminal DNA]. Zhonghua Nan Ke Xue. 2013 Jul;19(7):652-6. Chinese. PMID 23926686
- [Result] Brouillet S, Gala A, Barry F, Anav M, Ferrieres-Hoa A, Andreeva A, Molinari N, Gaspari L, Loup V, Anahory T, Hamamah S. Artificial shrinkage before fresh blastocyst transfer and IVF outcomes: a pilot randomized controlled study. Reprod Biomed Online. 2024 Aug;49(2):103941. doi: 10.1016/j.rbmo.2024.103941. Epub 2024 Mar 8. PMID 38824764